CLINICAL TRIAL: NCT07102225
Title: Effects of Intra-articular Hypertonic Dextrose and Hyaluronic Acid on Primary Knee Osteoarthritis: A Randomized Control Trial
Brief Title: Effects of Intra-articular Hypertonic Dextrose and Hyaluronic Acid on Primary Knee Osteoarthritis.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Raju Dey, Director, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5506
Record Dates: First submitted 2025-07-08; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Mild to Moderate Knee OA
MeSH Terms: interventions — Glucose; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of intra-articular hypertonic dextrose and hyaluronic acid on primary knee ostosteoarthritis (Experimental): To see the effectiveness of intra-articular hypertonic dextrose versus hyaluronic acid on primary knee OA
  Interventions: Drug: prolotherapy solution of 20% dextrose; Drug: Hyaluronic Acid (HA)

INTERVENTIONS:
Drug: prolotherapy solution of 20% dextrose — This intervention is open label. Both participants and investigator will know about the intervention. Participants are allocated according to simple randomization by lottery. Two groups with each contain 28 participants. One group will be given a mixture of intra-articular injection of 5.6 ml 25% dextrose and 1.4 ml 2% lignocaine to achieve a final concentration 20% dextrose with 0.4% lignocaine in the involved knee joint. Another group will be given 1.4 ml 2% lignocaine followed by 2 ml high molecular weight hyaluronic acid intra-articularly in the involved joint.
Drug: Hyaluronic Acid (HA) — This intervention is open label. Both participants and investigator will know about the intervention. Participants are allocated according to simple randomization by lottery. Two groups with each contain 28 participants. One group will be given a mixture of intra-articular injection of 5.6 ml 25% dextrose and 1.4 ml 2% lignocaine to achieve a final concentration 20% dextrose with 0.4% lignocaine in the involved knee joint. Another group will be given 1.4 ml 2% lignocaine followed by 2 ml high molecular weight hyaluronic acid intra-articularly in the involved joint.

SUMMARY:
The aim of this study is to compare the effectiveness of intra-articular hypertonic dextrose and hyaluronic acid in managing pain and improving function in patients with primary knee osteoarthritis (KOA). This study will guide us to treat primary KOA patients with dextrose prolotherapy instead of hyaluronic acid more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA diagnosis satisfying the American College of Rheumatology clinical and radiographic criteria, Kellgren-Lawrence grade of II and III determined by Postero-anterior knee radiograph.
* Participants will have the ability to undergo 3 months of follow-up
* Participants who will agree to avoid non-steroidal anti-inflammatory drugs during the research (acetaminophen will be prescribed for intractable pain)

Exclusion Criteria:

* Participants who will give a self-reported history of knee surgery, fracture, or infection.
* Kellgren-Lawrence grade IV KOA.
* Participants on anticoagulants.
* Participants who will have previous history of intra-articular knee injection of HA or prolotherapy within 6 months.
* Participants who have malignant disease or secondary KOA.
* Participants who will have a history of comorbid illness(es) like chronic heart failure, advanced COPD, end-stage renal failure, advanced liver disease and poorly controlled DM.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Outcome 1: " VAS score at week 1", Outcome 2: "VAS score at week 4", Outcome 3: "VAS score at week 12",
  VAS consisting of a 100mm long horizontal line, where 0 at one end indicates no pain and 100 at another end indicates worst pain. Number of participants will be assessed from baseline in pain scores on the Visual Analog Scale at 1, 4 and 12 weeks after treatment completion. Lower scores indicate better outcomes.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Outcome 1: " WOMAC score at week 1", Outcome 2: " WOMAC score at week 4", Outcome 3: " WOMAC score at week 12"
  WOMAC is a questionnaire consisting of 24 items organized into 3 subscales like pain, stiffness and physical function that is used in patients with knee osteoarthritis. Total score ranges from 0 to 96, with higher scores indicating worse symptoms. Number of participants will be assessed from baseline on the WOMAC Scale at 1, 4 and 12 weeks after treatment completion. Lower scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Farzana Khan Shoma, MBBS, FCPS, Study Director — Bangladesh Medical University (formerly known as Bangabandhu Sheikh Mujib Medical University)
Locations (1):
- Bangladesh Medical University (formerly known as Bangabandhu Sheikh Mujib Medical University), Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided